CLINICAL TRIAL: NCT03011229
Title: Endoscopic Ultrasound Fine Needle Biopsy of Submucosal Lesions of the GI Tract; Finding the Right Needle - A Randomized Study
Brief Title: Endoscopic Ultrasound (EUS) Fine Needle Biopsy (FNB) Submucosal Nodule
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow enrollment
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: Pro00077315
Record Dates: First submitted 2016-12-28; First posted 2017-01-05 (Estimated); Last update posted 2020-05-07 (Actual); Status verified 2020-05

CONDITIONS: GI Lesions

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Pro Core (Active Comparator): Subject is randomized to ProCore standard needle.
  Interventions: Device: Pro Core Needle
- Medtronic Shark Core (Experimental): Subject is randomized to Medtronic Sharkcore needle
  Interventions: Device: medtronic Sharkcore Needle

INTERVENTIONS:
Device: Pro Core Needle — Needle will be used in standard fashion utilizing a slow pull technique by an expert endoscopist who is familiar with EUS and use of both needles.
  Arms: Pro Core
Device: medtronic Sharkcore Needle — Needle will be used in standard fashion utilizing a slow pull technique by an expert endoscopist who is familiar with EUS and use of both needles.
  Arms: Medtronic Shark Core

SUMMARY:
The purpose of this study is to compare the diagnostic accuracy of a novel endoscopic ultrasound (EUS) biopsy needle to the current standard EUS needle.

The investigators hypothesize that with the SharkcoreTM needle a diagnostic yield of 90% is possible for subepithelial lesions (SEL) within the Gastrointestinal (GI) tract versus 60% yield with the current needle.

ELIGIBILITY:
Inclusion Criteria:

* Patients age 18 or older referred for EUS found to have a hypoechoic lesion > 8 mm within the GI lumen arising from the muscularis propria, as determined by EUS.
* Women that have a negative pregnant test

Exclusion Criteria:

* Patients under the age of 18.
* Uncorrectable coagulopathy (INR>1.5)
* Uncorrectable thrombocytopenia (platelet count <50,000)
* Patient who is unable to comply with study requirements
* Pregnant women
* Female patients who are not tested per our current unit protocol
* Refusal to consent or unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-09-05 (Actual); Primary Completion 2019-09 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
diagnostic accuracy of biopsy needle | end of biopsy, approximately 10 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Spaete, Principal Investigator — Duke Health System
Locations (1):
- Duke, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No